CLINICAL TRIAL: NCT00899223
Title: The CALGB Leukemia Tissue Bank
Brief Title: Collecting and Storing Blood, Bone Marrow, and Other Samples From Patients With Acute Leukemia, Chronic Leukemia, or Myelodysplastic Syndromes
Status: Active, not recruiting | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9665; U10CA031946 (NIH); CALGB-9665; CDR0000271412 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Leukemia; Chronic Leukemia; Myelodysplasia
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Bone Marrow Aspirate: 5 mL of bone marrow aspirate at the time of diagnosis, relapse, and during remission for each CALGB leukemia or myelodysplastic syndrome treatment protocol.
  * Blood: 10 mL of whole blood at the time of diagnosis, relapse, and during remission for each CALGB leukemia or myelodysplastic syndrome treatment protocol.
  * Buccal Cell Sample: One buccal cell sample at time of diagnosis, but may be obtained at other times if not done so previously

GROUPS / COHORTS (1):
- Group 1: Previously untreated patients on a CALGB treatment protocol for leukemia (acute or chronic) or myelodysplasia are eligible. Patients must be registered to CALGB 9665 prior to receiving any therapy for their disease.
  Interventions: Other: biologic sample preservation procedure

INTERVENTIONS:
Other: biologic sample preservation procedure

SUMMARY:
As one of the nation's largest cooperative cancer treatment groups, the Alliance for Clinical Trials in Oncology (Alliance) is in a unique position to organize a Leukemia Tissue Bank. The member institutions diagnose hundreds of patients with leukemia or myelodysplastic syndrome each year, and uniformly treat these patients with chemotherapy regimens. The Alliance offers centralized data management for the clinical history, the classification of the leukemia and myelodysplastic syndrome, cytogenetics, flow cytometric analysis, treatment and follow-up. The highly skilled health care providers at each member institution are familiar with obtaining informed consent, completing data questionnaires and shipping specimens. There currently exists a central processing facility where samples are prepared for a variety of cellular and molecular studies. Hence, the patient resources, the health care providers, and a processing facility for a Leukemia Tissue Bank are all in place. What is needed, however, and is addressed in the current protocol, is a formal mechanism to procure bone marrow, blood and normal tissue from patients with hematologic malignancies who are to be enrolled on Alliance (Cancer and Leukemia Group B [CALGB]) treatment studies.

DETAILED DESCRIPTION:
The objective of the study is to collect and store specimens from every newly diagnosed patient with acute or chronic leukemia or myelodysplastic syndrome (MDS) who are entered on a CALGB protocol for previously untreated patients. Bone marrow aspirate and blood specimens are obtained from patients at diagnosis, remission, or relapse and stored. Buccal smears are obtained at diagnosis, and DNA is extracted and preserved.

It was anticipated that the specimens collected under this protocol would be used by a large number of investigators. This protocol does not describe the details of each approved project (eg, eligibility age range).

ELIGIBILITY:
* Previously untreated patients on a CALGB treatment protocol for leukemia (acute or chronic) or myelodysplasia are eligible. Patients must be registered to CALGB 9665 prior to receiving any therapy for their disease.
* Signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with leukemia or myelodysplasia.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 1996-05 (Actual); Primary Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Collection and storage of specimens from newly diagnosed patients with acute or chronic leukemia or myelodysplastic syndromes enrolled on a CALGB protocol | At diagnosis
Collection and storage of specimens from newly diagnosed patients with acute or chronic leukemia or myelodysplastic syndromes enrolled on a CALGB protocol | At relapse
Collection and storage of specimens from newly diagnosed patients with acute or chronic leukemia or myelodysplastic syndromes enrolled on a CALGB protocol | At remission

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caligiuri, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (142):
- United States (142):
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Pismo Beach, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Cleveland Regional Medical Center, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - McLeod Regional Medical Center, Florence, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Liu TH, Raval A, Chen SS, Matkovic JJ, Byrd JC, Plass C. CpG island methylation and expression of the secreted frizzled-related protein gene family in chronic lymphocytic leukemia. Cancer Res. 2006 Jan 15;66(2):653-8. doi: 10.1158/0008-5472.CAN-05-3712. PMID 16423993
- [Derived] Archer KJ, Fu H, Mrozek K, Nicolet D, Mims AS, Uy GL, Stock W, Byrd JC, Hiddemann W, Braess J, Spiekermann K, Metzeler KH, Herold T, Eisfeld AK. Identifying long-term survivors and those at higher or lower risk of relapse among patients with cytogenetically normal acute myeloid leukemia using a high-dimensional mixture cure model. J Hematol Oncol. 2024 May 3;17(1):28. doi: 10.1186/s13045-024-01553-6. PMID 38702786
- [Derived] Ozga M, Nicolet D, Mrozek K, Yilmaz AS, Kohlschmidt J, Larkin KT, Blachly JS, Oakes CC, Buss J, Walker CJ, Orwick S, Jurinovic V, Rothenberg-Thurley M, Dufour A, Schneider S, Sauerland MC, Gorlich D, Krug U, Berdel WE, Woermann BJ, Hiddemann W, Braess J, Subklewe M, Spiekermann K, Carroll AJ, Blum WG, Powell BL, Kolitz JE, Moore JO, Mayer RJ, Larson RA, Uy GL, Stock W, Metzeler KH, Grimes HL, Byrd JC, Salomonis N, Herold T, Mims AS, Eisfeld AK. Sex-associated differences in frequencies and prognostic impact of recurrent genetic alterations in adult acute myeloid leukemia (Alliance, AMLCG). Leukemia. 2024 Jan;38(1):45-57. doi: 10.1038/s41375-023-02068-8. Epub 2023 Nov 28. PMID 38017103
- [Derived] Rebechi M, Kohlschmidt J, Mrozek K, Nicolet D, Mims AS, Blachly JS, Orwick S, Larkin KT, Oakes CC, Hantel A, Carroll AJ, Blum WG, Powell BL, Uy GL, Stone RM, Larson RA, Byrd JC, Paskett ED, Plascak JJ, Eisfeld AK. Association of social deprivation with survival in younger adult patients with AML: an Alliance study. Blood Adv. 2023 Aug 8;7(15):4019-4023. doi: 10.1182/bloodadvances.2022009325. No abstract available. PMID 37196637
- [Derived] Mrozek K, Kohlschmidt J, Blachly JS, Nicolet D, Carroll AJ, Archer KJ, Mims AS, Larkin KT, Orwick S, Oakes CC, Kolitz JE, Powell BL, Blum WG, Marcucci G, Baer MR, Uy GL, Stock W, Byrd JC, Eisfeld AK. Outcome prediction by the 2022 European LeukemiaNet genetic-risk classification for adults with acute myeloid leukemia: an Alliance study. Leukemia. 2023 Apr;37(4):788-798. doi: 10.1038/s41375-023-01846-8. Epub 2023 Feb 23. PMID 36823396
- [Derived] Fobare S, Kohlschmidt J, Ozer HG, Mrozek K, Nicolet D, Mims AS, Garzon R, Blachly JS, Orwick S, Carroll AJ, Stone RM, Wang ES, Kolitz JE, Powell BL, Oakes CC, Eisfeld AK, Hertlein E, Byrd JC. Molecular, clinical, and prognostic implications of PTPN11 mutations in acute myeloid leukemia. Blood Adv. 2022 Mar 8;6(5):1371-1380. doi: 10.1182/bloodadvances.2021006242. PMID 34847232
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516